CLINICAL TRIAL: NCT07161583
Title: Post-Market Clinical Follow-up Registry to Evaluate the Safety and Performance of the Atrium Advanta VXT and Flixene Vascular Grafts in Patients Undergoing Surgical Repair or Replacement of Peripheral Arteries
Brief Title: Advanta VXT and Flixene PMCF Registry
Status: Recruiting | Type: Observational
Sponsor: Atrium Medical Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: DD021215-001
Record Dates: First submitted 2025-08-12; First posted 2025-09-08 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Peripheral Arterial Disease (PAD) Cohort
  Interventions: Device: Advanta VXT Vascular Graft; Device: Flixene Vascular Graft

INTERVENTIONS:
Device: Advanta VXT Vascular Graft — The Advanta VXT graft is a two (2)-layer graft employing a single layer ePTFE graft, which is then wrapped with an additional layer of ePTFE for increased support. Some Advanta VXT configurations include Helix, which is a monofilament bead wrapped circumferentially around a portion or the entire length of the graft (such a graft is also called a Ringed Graft). The helix rings are bonded to the exterior surface of the graft. Advanta VXT Tapers are formed by changing the graft diameter, expanding from a small Inner Diameter (ID) to a larger ID (with the result that one end is larger).
Device: Flixene Vascular Graft — The Flixene vascular graft is a three (3)-layered graft comprised of ePTFE. The Flixene graft was designed with an additional layer of ePTFE. As a result of its design, ring support is not necessary

SUMMARY:
The purpose of the registry is to evaluate the long-term safety and performance of Advanta VXT and Flixene vascular grafts for repair or replacement of peripheral arteries. This registry is also intended to provide further data on the clinical usefulness of the Advanta VXT and Flixene vascular grafts.

ELIGIBILITY:
Inclusion Criteria:

* Willing, and able to provide legally-effective written informed consent (as required by IRB/EC)
* Male and female patients that have undergone replacement or repair of the peripheral arteries using the Advanta VXT or Flixene vascular graft.
* Were at least 18 years of age at the time of the procedure
* Available records for data collection, with a minimum of 36 months of data/follow-up.

Exclusion Criteria:

- Active infection in the region of graft placement at the time of implantation of the Advanta VXT or Flixene vascular graft

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: An approximate 1,000 patients from 25 sites across the US and Europe will participate in this registry. The number of patients and sites included will ensure a representation of the overall population, specifically in vascular surgery. No mandated procedures, assessments or visits will be implemented, given the non-interventional nature of the registry.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-09-25 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants meeting Primary Efficacy Endpoint | Procedure/surgery through registry completion (a minimum of 3 years)
  Primary patency defined as freedom from graft occlusion or reintervention
Percentage of Participants meeting Primary Safety Endpoint | Procedure/surgery through registry completion (a minimum of 3 years)
  Major Adverse Limb Events (MALE), defined as major amputation or major reintervention, including placement of a new bypass graft, interposition graft, thrombectomy, or thrombolysis

SECONDARY OUTCOMES:
Incidence of Reported Complications/Events | Procedure/surgery through registry completion (a minimum of 3 years)
Percentage of Participants meeting Primary-Assisted Graft Patency | Procedure/surgery through registry completion (a minimum of 3 years)
  Defined as freedom from graft occlusion irrespective of whether an intervention was performed; in other words, primary-assisted patency is not lost when a reintervention is performed to preserve graft patency before occlusion occurs
Percentage of Participants meeting Secondary Graft Patency | Procedure/surgery through registry completion (a minimum of 3 years)
  Defined as freedom from "permanent" loss of graft patency
Rate of change in Rutherford Category | Baseline, procedure/surgery, through registry completion (a minimum of 3 years)
Rate of change in Ankle-Brachial Index (ABI) | Baseline, procedure/surgery, through registry completion (a minimum of 3 years)

CONTACTS AND LOCATIONS:
Overall Officials: Director, Clinical Affairs, Study Director — Getinge
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No